CLINICAL TRIAL: NCT06936150
Title: Effect of Tourniquet Use on Index of Cardiac-Electrophysiological Balance Calculations (ICEB and ICEBc) in Upper Extremity Surgeries
Brief Title: Effect of Tourniquet Use on ICEB and ICEBc in Upper Extremity Surgeries
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Fatma Nur Arslan, MD, Anesthesiology and Reanimation, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-13/108
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Arrhythmia, Cardiac; Tourniquet Complications
Keywords: ICEB; ICEBc; Surgical Tourniquet; Cardiac Arrhytmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Electrocardiography — Electrocardiography (ECG) is a non-invasive test used to measure the electrical activity of the heart. It involves placing electrodes on all four extremities and the chest area of the person and measuring the derivation between these electrodes. This procedure is painless and does not contain any elements that will disrupt the integrity of the body.

SUMMARY:
In our study, we will examine whether the pressure bandage (tourniquet) used to reduce bleeding during surgery in patients with arm fractures has an effect on heart rhythm. Tourniquet use is routinely used in every patient in these surgeries. This procedure reduces blood flow to the area where the surgery will be performed by applying a pressure bandage in order to reduce bleeding. At the end of the surgery, this bandage is removed and the blood flow returns to normal. Blood pressure changes that may occur during this process and the cellular effects of the changing blood flow may cause some changes in heart rhythm.

To observe those changes, during the operation, an electrocardiogram (ECG, heart graph) will be taken to determine changes in heart rhythm before and after the tourniquet is applied. An ECG is also performed before the surgery for preoperative anesthesia evaluation. The ECG procedure is a painless procedure that takes about 1 minute, includes placing probes on the chest and does not disrupt the integrity of the skin..The procedure will be performed while patients are under anesthesia.

Calculations will be made by the parameters on the ECG. Apart from taking an ECG, no other procedure will be performed on the patients

DETAILED DESCRIPTION:
The use of a tourniquet during surgical repair of traumatic upper extremity fractures is a very common practice. Surgical Tourniquets are used in orthopaedic for creation of a bloodless field, greater safety, better precision, and more convenience for the surgeon. Despite the ease it provides in terms of surgery, the use of a tourniquet can lead to some complications.

Most surgical tourniquets are of the pneumatic design.(1) When using a pneumatic tourniquet in upper extremity surgeries, a pressure of 150-250 mmHg is usually applied. The blood flow to the extremity is cut off by this pressure effect. However, stopping the circulation causes temporary ischemia. Limb occlusion causes metabolic changes in the ischemic limb that include: Increased lactic acid, PaCO2 and potassium levels, and decreased levels of PaO2, and pH. Toxic metabolites produce pathophysiological changes when released into the general circulation.(2, 3). The degree of these changes correlates with the duration of ischemia. All of these changes are fully reversed within 30 min of tourniquet deflation. (4) These metabolic changes may have negative effects on cardiac electrical activity. Theoretically, there is a risk that these ischemic metabolites and pH changes may trigger cardiac arrhythmias.

Indeed, pre-clinical studies demonstrated that λ,( λ=effective refractory period × conduction velocity) was the best predictor of arrhythmic tendency, increasing with pro-arrhythmic conditions and decreasing by anti-arrhythmic therapy.(5) The fact that λ must be assessed invasively using electrophysiological investigations in a clinical context is a significant drawback, though. The index of Cardiac-Electrophysiological Balance" (iCEB), which is the ratio of QT/QRS of the ECG, was proposed as the noninvasively measured equivalent of λ by Lu et al.(6) In addition, ICEBc, a version calculated with Qtc instead of Qt, has been used in various studies to predict arrhythmia risk, similar to ICEB (7, 8).

In our study, we aimed to investigate whether ischemic metabolites and other systemic effects occurring after tourniquet application in upper extremity surgeries create any changes on the ICEB and ICEBc values of patients.

The study was designed as a prospective, observational study. Patients were included in the study after their consent to participate was obtained by the anesthesiologists during the preoperative evaluation in the anesthesia outpatient clinic of a training and research hospital. All data related to the study were recorded by the same anesthesia team.

During the preoperative evaluation, American Society of Anesthesiology (ASA) risk group I-III, patients between the ages of 18-65, who were scheduled for elective upper extremity fixation surgery were included in the study.

Patients with bundle branch block in preoperative ECG, patients with arrhythmia, those taking antiarrhythmic drugs, those with pacemakers, patients with known drug-specific allergies, and patients with electrolyte disorders were not included in the study.

The primary outcome of our study was whether there was a significant increase in ICEB and ICEBc values after tourniquet deflation compared to before opening. The secondary outcome of the study was whether there was a significant increase in ICEB and ICEBc values measured at the beginning and end of surgery.

For upper extremity fixation surgery, before anesthesia induction (ICEB1/ICEBc1), after induction (ICEB2/ICEBc2), 5 minutes before the tourniquet was inflated (ICEB3/ICEBc3), 5 minutes after it was inflated (ICEB4/ICEBc4), 5 minutes before the tourniquet was opened (ICEB5/ICEBc5) and 5 minutes after it was opened (ICEB6/ICEBc6), ECG was taken . ECG measurements were performed and ICEB and ICEBc values were calculated using the D II and V5 derivations in these ECGs. After calculating QT, QTc and QRS durations, iCEB and ICEBc calculations will be made. iCEB is calculated by dividing the QT interval by the QRS duration (QT/ QRS). iCEBc is calculated by dividing the QTc interval by the QRS duration (QTc/ QRS).

Simultaneously, mean arterial pressure, heart rate, oxygen saturation were recorded non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) risk group I-III, patients
* Upper extremity fracture which requires tourniquet application during surgery

Exclusion Criteria:

* bundle branch block in preoperative ECG
* patients with arrhythmia
* those taking antiarrhythmic drugs
* those with pacemakers
* patients with known drug-specific allergies
* patients with electrolyte disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients who applied to the orthopedics and traumatology department of the training and research hospital due to isolated fractures in the upper extremity and were planned for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Change of ICEB and ICEBc with the opening of the tourniquet | Difference between 5 minutes before the end of the surgical tourniquet application and 5 minutes after the tourniquet was opened
  Primary outcome is whether there was a significant increase in ICEB and ICEBc values after tourniquet deflation compared to before opening

SECONDARY OUTCOMES:
Changes in ICEB and ICEBc during surgery | The time interval between the minute immediately before the start of anesthesia and 5 minutes after the tourniquet is opened.
  The secondary outcome of the study was whether there was a significant increase in ICEB and ICEBc values measured at the beginning and end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Research and Education Hospital, Kırşehir/Merkez, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided whether to share the IPDs of our study.